CLINICAL TRIAL: NCT05418231
Title: Observation of the Natural Course of Dry Age-related Macular Degeneration
Brief Title: Observation of the Natural Course of Age-related Macular Degeneration
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SXD20220609
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Dry Age-related Macular Degeneration; Macular Degeneration, Dry
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research will study natural course of dry AMD in Chinese population, screen fundus imaging indicators for patients with Chinese dry AMD, describe the clinical features of Chinese patients with dry AMD, and obtain a biological sample library of dry AMD mainly in China.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 yrs male or female AMD patients
* Dry-AMD patients in either early, intermediate, or intermediate-to-late stage confirmed by fundus examinations.

Exclusion Criteria:

* Any eye with disease that would interfere with the retinal examinations
* Research eye with CNV or high myopia
* Surgeries that may interfere with AMD evaluation
* Long-term uses of medications that are associated with retinal or neural toxicities.
* IOP more than 26 mmHg
* Received cataract surgery in 3 months.
* Other conditions: diseases that causes less than 5 years survival; any condition that causes high risk of drop-out, or low compliance, for instance cognition disorder; have been involved in other trial that interfere with the current visit plan; taking other angiogenesis Inhibitors drugs for treating cancer.
* Other conditions not suitable for the current study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dry AMD patients in Shanghai General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 60 months
  A typical ETDRS chart that if frequently used for visual acuity testing

SECONDARY OUTCOMES:
Drusen density and shape | 60 months
  Drusen Measurement on OCT or Fundus photography
The rate of 5-year progression | 60 months
  The evaluation criteria for progression: progress to intermediate (only for patients with early phase AMD at baseline) or intermediate-to-late, or late stage AMD.
GA growth rate | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, PHD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided